CLINICAL TRIAL: NCT05674331
Title: Clinical, Radiographical, Histological Evaluation and Blood Flow Analysis of Hard- and Soft- Tissue Changes Following Alveolar Ridge Preservation
Brief Title: Clinical, Radiographical, Histological Evaluation and Blood Flow Analysis of Alveolar Ridge Preservation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Eleonora Solyom, PhD student, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARP-Semmelweis-Paro
Record Dates: First submitted 2022-11-16; First posted 2023-01-06 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Alveolar Bone Loss
Keywords: alveolar ridge preservation; autogenous tooth bone graft; extraction side development technique
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- socket seal group (Active Comparator): After tooth extraction a soft tissue pounch is sutured above the extraction socket.
  Interventions: Procedure: Socket seal technique
- XSD+ socket seal group (Experimental): After tooth extraction for the reconstruction of the buccal bony wall a xenograft membrane with a long absorption rate is fixed with titanium pins to the buccal side. A soft tissue pounch is sutured above the extraction socket.
  Interventions: Procedure: Extraction site development technique; Procedure: Socket seal technique
- XSD+ ATB+socket seal group (Experimental): After tooth extraction, the tooth will be grinded and after the sterilization procedure it will be filled back to the extraction socket. For the reconstruction of the buccal bony wall a xenograft membrane with a long absorption rate is fixed with titanium pins to the buccal side. A soft tissue pounch is sutured above the extraction socket.
  Interventions: Procedure: Extraction site development technique; Device: autogenous tooth bone graft; Procedure: Socket seal technique

INTERVENTIONS:
Procedure: Extraction site development technique — The technique is described by Molnar et al. in 2019. The aim is to reconstruct the buccal bony wall with a xenogenic membrane with a slow absorption rate properties. This technique aims to stabilizate and enlarge the blood clot .
  Other Names: XSD
  Arms: XSD+ ATB+socket seal group; XSD+ socket seal group
Device: autogenous tooth bone graft — ATB was invented by Kim et al. in 2011. The extracted tooth is grinded and goes throw a sterilization procedure by the manufacturer's recommendation. The graft material can be used immediately for ARP.
  Other Names: ATB
  Arms: XSD+ ATB+socket seal group
Procedure: Socket seal technique — After tooth removal neither graft nor any membrane material is inserted to the extraction socket. A soft tissue pounch is harvested from the hard palate and it is fixed above the extraction socket with single interrupted sutures.

SUMMARY:
With alveolar ridge preservation (ARP) ridge resorption following extraction may be reduced. Several materials and techniques have been advocated for ARP. The aim of our randomised clinical trial is to evaluate the efficacy of extraction side development technique (XSD) and autogenous tooth bone graft (ATB) for ARP.

DETAILED DESCRIPTION:
A three armed clinical study will be established. According to the sample size calculation, every arm will contain 21 participants. The first group is the socket seal group. In the second group we aim to combine the socket seal and XSD technique. In the third group the XSD technique will be combined with the ATB material. The primary outcome is the alveolar ridge width change in millimeter, measured immediately after the tooth extraction and after 6 months at the reentry procedure. The change in alveolar ridge width and vertical dimensional alterations will be also measured as secondary outcomes on the CBCT at baseline and after 6 months. Further secondary outcomes are the monitoring of gingival microvascularization, monitoring of flap revascularization by Laser Speckle Contrast Imaging and assessment of soft tissue volumetric changes by intraoral scanning and histomorphometric evaluation of the volumetric percentage of newly formed bone, connective tissue and graft material after a 6-month healing period in a core biopsy taken at the time of implant placement.

Hypothesis: The XSD and XSD+ATB groups are expected to have less pronounced horizontal width losses. XSD group is expected to produce the highest graft turnover.

ELIGIBILITY:
Inclusion Criteria:

* Women and men Patients over 18 years Co-operative patients with good individual oral hygiene (FMBS: 25%>) Patients with periodontal disease in treatment or under treatment with minimal active inflammation (FMPS: 25%>)

Local criteria:

Teeth with a hopeless prognosis with advanced periodontal or endo-periodontal defects, which are restored with implant prosthesis EDS 3-4 extraction defects after tooth extraction

Exclusion Criteria:

* Infectious diseases (HBV, HCV, HIV, CoV-2019…) Current chemotherapy or radiotherapy Previous radiation therapy to the head and neck region (in the last 2 years) Untreated insulin dependent diabetes mellitus Clinically significant osteoporosis or other systemic disease affecting bone metabolism Clinically significant circulatory disorder e.g.: decompensated cardiac failure Haemodynamically significant valvular heart failure or myocardial infarction within the last 3 months Clinically significant coagulopathy Current or previous systemic corticosteroid therapy (in the last 2 months) Current or previous systemic bisphosphonate therapy (beyond 30 days) Pregnant or breastfeeding women Smoking (max 5 cigarettes per day) Drug addiction, alcoholism

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Horizontal ridge width changes | during first surgery and during 6 months reentry
  The primary outcome is the alveolar ridge width change in millimeter intraoperatively, measured immediately after the tooth extraction and after 6 months at the reentry procedure (at the time of implant placement).

SECONDARY OUTCOMES:
Evaluation of change of alveolar ridge width on CBCT | at baseline and 6 months postoperatively
  Alveolar ridge width measured at baseline and 6 months postoperatively on CBCT data sets
Evaluation of change of alveolar ridge height on CBCT | at baseline and 6 months postoperatively
  Alveolar ridge height measured at baseline and 6 months postoperatively on CBCT data sets
Evaluation of change of alveolar ridge volume on CBCT | at baseline and 6 months postoperatively
  Alveolar ridge volumetric changes measured at baseline and 6 months postoperatively on CBCT data sets
Monitoring the microvascularization | Pre-operative and 1, 3, 5, 7, 10, 14, 21, 28 days and 2, 3, 4, 5 and 6 months after surgeries.
  Monitoring of gingival microvascularization, monitoring of flap revascularization by Laser Speckle Contrast Imaging
Examination of early wound healing phase | Pre-operative and 1, 3, 5, 7, 10, 14, 21, 28 days and 2, 3, 4, 5 and 6 months after surgeries.
  Examination of early wound healing phase by means of clinical photdocumentation
Soft tissue volumetric changes | analysis of baseline and 6-month post-alveolar digital impressions
  Assessment of soft tissue volumetric changes by intraoral scanning
Histomorphometry | 6 months postoperatively
  Histomorphometric evaluation of the volumetric percentage of newly formed bone, connective tissue and graft material after a 6-month healing period in a core biopsy taken at the time of implant placement

CONTACTS AND LOCATIONS:
Overall Officials: Balint Molnar, Principal Investigator — Department of Periodontology,Semmelweis University
Locations (1):
- Semmelweis University Department of Periodontology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No